CLINICAL TRIAL: NCT00625118
Title: A Study to Gather Safety Data Following Administration of a Hib-containing Booster Vaccine in Children Aged Two to Five Years
Acronym: DIPS
Status: Completed | Type: Observational
Sponsor: Public Health England (Other Government)
Responsible Party: Prof Elizabeth Miller, Health Protection Agency
Other Study IDs: DIPS
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2009-01

CONDITIONS: Haemophilus Infections
Keywords: Hib conjugate vaccine; reactogenicity; local reactions; systemic symptoms
MeSH Terms: conditions — Haemophilus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Children in receipt of a Hib containing vaccine at pre-school booster (3.5-6 years old).

SUMMARY:
This will be an observational study where parents/ guardians of children in receipt of their preschool booster will be approached for their child(ren) to take part. Following written informed consent the Vaccine Research Nurse will explain the purpose of the study and what would be involved. Participation will involve completion of a health diary for the week following vaccination to document how their child has been both in terms of local reactions and systemic symptoms as well as any visits to a doctor (GP or hospital). The nurse will telephone the family at 48-72 hours following vaccination to see how the child has been. Information about the vaccine given in the current campaign and vaccines administered in the infant schedule including date of administration, product and batch number will be recorded where available.

Should any large local reactions be reported the nurse may visit the child to take a photograph to document and illustrate these - photographs will be taken without the child's face visible.

Subjects will be recruited in two centres - Hertfordshire and Gloucestershire. Recruitment will start as soon as the necessary approvals are in place. Monthly reports of observed data will be submitted to the MHRA though the formal analysis will not be conducted until the end of the study.

Recruitment figures and the incidence of ESLs will be reviewed on a six-monthly basis.

At this point it is difficult to predict parental attitude to taking part, though from experience with recruitment in previous studies it is hoped this will be positive, so affording a large number of participants.

DETAILED DESCRIPTION:
Medicines, including vaccines, are monitored by the Medicines and Healthcare Regulatory Agency (MHRA) using what is commonly known as the "yellow card system" where patients or healthcare professionals may submit notifications. This involves reporting any untoward medical event that it is suspected may be related to administration of the given medicine. Through this system concern has been raised about large local reactions, particularly extensive limb swelling (ESL) which is usually defined as an area more than or equal to 50mm, in young children in receipt of their pre-school booster. The preschool booster vaccine contains diphtheria (D), tetanus (T), pertussis (P) and inactivated polio vaccine (IPV). Most of the children about whom these yellow card safety reports have been submitted would have been primed with whole cell pertussis (wP) containing vaccines in infancy. In some cases reports have noted blistering and cellulitis in the vaccinated limb with antibiotic treatment prescribed. There is a recognised risk of ESL in a small proportion of children, 2-13%, following administration of a fourth or fifth dose of acellular-pertussis containing vaccine. In previous studies these local reactions fully resolved without treatment within a few days. Acellular pertussis (aP) containing vaccine has been used exclusively in the routine infant immunisation programme in teh UK since September 2004. The first children who received a primary immunisation course exclusively of aP containing vaccine will reach 3.5 years, the age at which their preschool booster will be given, from December 2007. This will be their fourth dose of the aP containing vaccine and therefore provides the opportunity to define with greater precision the incidence of ESL following vaccination in UK children with regard to primary immunisation history of aP vs the previously used whole cell pertussis (wP) vaccines. These children have been subject to a unique vaccination schedule compared to those in the previous studies mentioned above. They will have been vaccinated under an accelerated schedule compared to most other countries, at 2, 3 and 4 months, and will have had meningococcal conjugate vaccine at the same time as their other primary immunisations. To that end we will be asking parents/ guardians of individuals in receipt of the pre-school booster to complete a health diary for a week following vaccination.

Changes to the routine pre-school booster have recently been announced. These have been instituted to provide a fourth dose of Hib vaccine to a cohort of children who, by virtue of their birth date, have not had this dose. The lack of a fourth dose of Hib vaccine has been recognised by the UK Department of Health Joint Committee for Vaccination and Immunisation as potentially putting this group of children at greater risk of Hib disease. These children have birth dates between 13 March 2003 and 3 September 2005 and were too young to be included in the Hib catch up campaign in 2004, which included all children born April 1999 to October 2002 (ie 6 months to 4 years at the start of the campaign) and all those becoming 6 months of age during the campaign (ie born October 2002 to March 2003) and are too old to have received a dose of Menitorix since its introduction to the national schedule in September 2006. The objective of the recently announced programme is to deliver a safe and effective booster vaccine in the most logistically simple and cost-effective way. To that end most eligible children will be given the Hib vaccine alongside the routine pre-school booster. At pre-school, children are vaccinated with DTaP and inactivated polio vaccine (IPV). The Hib vaccine will be delivered in the form of Infanrix-IPV-Hib or Pediacel which are both DTaP-Hib-IPV combinations. There is a small percentage of children identified who have already had their pre-school booster without the Hib component, so they will be re-called and offered a dose of Menitorix, the MenC and Hib conjugate vaccine. The vaccines to be used in this Hib campaign may be given to some children above the upper age limit specified in their Summary of Product Characteristics (SPC) and in addition differ in antigen content from those normally given at this age:

* Pediacel contains higher doses of diphtheria and some of the acellular pertussis components than Repevax. The diphtheria content has previously been shown not to affect reactogenicity as has the aP with the exception of swelling =3 cms on day 2 after vaccination where swelling >=3cm occurred in 17.5% of DTaP recipients compared with 10.0% of DT recipients (p= 0.02).
* Older children will receive the tetanus conjugated Menitorix only a month after receipt of their pre-school booster and may therefore have high tetanus antibody levels. This has previously been shown to have no association with reactogenicity in a study where the tetanus conjugate dose was similar to that included in the Menitorix vaccine. One of the main objectives of the UK Vaccine Evaluation Consortium is to provide data that can be used in planning and refining the national immunisation programme. Though there is a body of evidence to support the safety of this campaign, it nevertheless provides a natural opportunity for specialist Vaccine Research Nurses to interact with parents in collecting safety data following administration of the preschool booster.

ELIGIBILITY:
Inclusion Criteria:

* Child in receipt of the preschool booster vaccination or Menitorix under the Hib catchup campaign
* Written informed consent from a parent/ guardian

Exclusion Criteria:

* None

Ages: 42 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children in receipt of pre-school booster vaccinations (age 3.5-6 years)
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MB BS FFPHM FRCPath, Principal Investigator — Public Health England
Locations (2):
- United Kingdom (2):
  - Health Protection Agency, Gloucester
  - Health Protection Agency, London

REFERENCES:
- [Background] Southern J, Waight PA, Andrews N, Miller E. Extensive swelling of the limb and systemic symptoms after a fourth dose of acellular pertussis containing vaccines in England in children aged 3-6years. Vaccine. 2017 Jan 23;35(4):619-625. doi: 10.1016/j.vaccine.2016.12.017. Epub 2016 Dec 23. PMID 28017441
- See also: Published study results — https://www.ncbi.nlm.nih.gov/pubmed/28017441